CLINICAL TRIAL: NCT06622395
Title: Telepsychiatry in Children: Diagnostic Evaluation of Autism Spectrum Disorder
Acronym: TELE-TSA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier St Anne (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: D21-P021; IDRCB:2021-A02675-36 (Other: GHU Paris)
Record Dates: First submitted 2024-09-26; First posted 2024-10-02 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Autism Spectrum Disorder (ASD); Neurodevelopmental Disorders
Keywords: Telepsychiatry; Remote Diagnosis; Autism Diagnosis; ADOS-2; BOSA; ADI-R; Teleconsultation; Pediatric ASD Diagnosis
MeSH Terms: conditions — Autism Spectrum Disorder; Neurodevelopmental Disorders

STUDY DESIGN:
Intervention Model Description: This is a prospective, single-center study aimed at testing the validity of the remote diagnostic modality for patients aged 24 months to 5 years with neurodevelopmental disorders (NDD) and suspected Autism Spectrum Disorder (ASD), involving second or third-line professional intervention. The study is designed sequentially in groups using the Fleming model (Group-Sequential Tests for One Proportion in a Fleming Design). The adopted model includes two interim stages.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remote Diagnosis Arm (Experimental): Remote Diagnostic Arm (Teleconsultation):
  First Teleconsultation (V1): A child psychiatrist or psychologist specializing in ASD conducts the ADI-R (short version) interview with the parents or legal guardian via teleconsultation. The professional will score the items from the algorithm. After the consultation, the professional completes a questionnaire assessing the technical aspects of the remote interview (e.g., video quality, connection stability).
  Second Teleconsultation (V2): During the BOSA remote assessment, the professional sends the parent/caregiver instructions and a video link. The parent watches the video and follows guidance on how to position themselves and the child for optimal visibility. The parent then carries out the BOSA activities under supervision. The professional observes the child's behavior and provides time guidance. Two questionnaires are completed: one on the technical aspects of the consultation and the second on parent-child interaction.
  Interventions: Diagnostic Test: Remote diagnosys
- In person Arm (No Intervention): In-person Arm (as usual) :
  Visit V0 (In-person ADI-R): The ADI-R interview is conducted in person by a psychiatrist or psychologist.
  Visit V3 (In-person ADOS-2): A different randomly assigned professional will perform an in-person ADOS-2 evaluation.

INTERVENTIONS:
Diagnostic Test: Remote diagnosys — Remote Diagnostic Arm (Teleconsultation): First Teleconsultation (V1): A child psychiatrist or psychologist specializing in ASD conducts the ADI-R (short version) interview with the parents or legal guardian via teleconsultation. The professional will score the items from the algorithm. After the consultation, the professional completes a questionnaire assessing the technical aspects of the remote interview (e.g., video quality, connection stability). Second Teleconsultation (V2): During the BOSA remote assessment, the professional sends the parent/caregiver instructions and a video link. The parent watches the video and follows guidance on how to position themselves and the child for optimal visibility. The parent then carries out the BOSA activities under supervision. The professional observes the child's behavior and provides time guidance. Two questionnaires are completed: one on the technical aspects of the consultation and the second on parent-child interaction.
  Arms: Remote Diagnosis Arm

SUMMARY:
Autism Spectrum Disorder (ASD) is a neurodevelopmental disorder recognized as a major national cause in 2012. The French Autism Plan 2018-2022 emphasizes early diagnosis and intervention for better cognitive and behavioral outcomes. The COVID-19 pandemic complicates the use of the ADOS-2 diagnostic tool due to mask-wearing and distancing requirements. To address this, the Brief Observation Symptoms of Autism (BOSA) has been adapted for remote assessment. The BOSA, translated into French, is recommended alongside the Autism Diagnostic Interview -Revised (ADI-R) for complementary diagnostic algorithms. No similar projects have been undertaken in France or Canada.

DETAILED DESCRIPTION:
Autism Spectrum Disorder (ASD) is a neurodevelopmental condition characterized by difficulties in social interaction, communication, and restricted, repetitive behaviors. Early diagnosis is critical for intervention and improving developmental outcomes. The French 2018-2022 Autism Plan emphasizes timely diagnosis to optimize care and reduce long-term impacts. Current tools, including the Autism Diagnostic Observation Schedule (ADOS-2) and the Autism Diagnostic Interview-Revised (ADI-R), are widely used but require in-person assessment. The COVID-19 pandemic has complicated the use of such tools due to mask-wearing and social distancing, limiting effective evaluation.

To address this, the Brief Observation of Symptoms of Autism (BOSA) has been adapted for remote use, offering a new approach to diagnosing ASD in children. This study will implement a teleconsultation model, utilizing BOSA and a shortened version of ADI-R, for children aged 24 months to 5 years with suspected ASD. The BOSA was adapted and translated into French under the approval of its creators and WPS publishing. The study aims to determine whether teleconsultation-based evaluations can achieve similar diagnostic accuracy as in-person assessments.

It is hypothesized that remote diagnosis using BOSA and ADI-R will have an accuracy rate of at least 80% compared to in-person ADOS-2 assessments, across key diagnostic domains such as social interaction, communication, and restrictive behaviors. The teleconsultation process may provide a more accessible, less disruptive diagnostic pathway, especially in situations where in-person evaluations are delayed or impractical.

This study will be one of the first in France and Canada to implement such a remote diagnostic model, addressing a gap in the literature and offering a potential solution to diagnostic delays caused by the pandemic. Concordance between teleconsultation and in-person diagnostic outcomes will be measured to assess the reliability and feasibility of this approach.

Autism Spectrum Disorder (ASD) is a neurodevelopmental condition characterized by difficulties in social interaction, communication, and restricted, repetitive behaviors. Early diagnosis is critical for intervention and improving developmental outcomes. The French 2018-2022 Autism Plan emphasizes timely diagnosis to optimize care and reduce long-term impacts. Current tools, including the Autism Diagnostic Observation Schedule (ADOS-2) and the Autism Diagnostic Interview-Revised (ADI-R), are widely used but require in-person assessment. The COVID-19 pandemic has complicated the use of such tools due to mask-wearing and social distancing, limiting effective evaluation.

To address this, the Brief Observation of Symptoms of Autism (BOSA) has been adapted for remote use, offering a new approach to diagnosing ASD in children. This study will implement a teleconsultation model, utilizing BOSA and a shortened version of ADI-R, for children aged 24 months to 5 years with suspected ASD. The BOSA was adapted and translated into French under the approval of its creators and WPS publishing. The study aims to determine whether teleconsultation-based evaluations can achieve similar diagnostic accuracy as in-person assessments.

It is hypothesized that remote diagnosis using BOSA and ADI-R will have an accuracy rate of at least 80% compared to in-person ADOS-2 assessments, across key diagnostic domains such as social interaction, communication, and restrictive behaviors. The teleconsultation process may provide a more accessible, less disruptive diagnostic pathway, especially in situations where in-person evaluations are delayed or impractical.

This study will be one of the first in France and Canada to implement such a remote diagnostic model, addressing a gap in the literature and offering a potential solution to diagnostic delays caused by the pandemic. Concordance between teleconsultation and in-person diagnostic outcomes will be measured to assess the reliability and feasibility of this approach.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 24 months to 5 years whose families request a diagnostic evaluation at the Autism and Related Disorders Research and Diagnostic Center (CREDAT).
* Consent to participate in the research in addition to their planned evaluation at the Autism and Related Disorders Research and Diagnostic Center (CREDAT), including consent collection procedures for minors.
* Sufficient understanding of the French language to complete the short version of the Autism Diagnostic Interview-Revised (ADI-R) and the Brief Observation of Symptoms of Autism (BOSA) assessment.

Exclusion Criteria:

* Lack of access to sufficient technology to participate in the protocol (teleconsultation).
* Refusal to participate in the research.
* Confirmed sensory or motor disorders (hearing or vision) that are not compensated (e.g., no glasses or hearing aids).

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 137 (Estimated)
Dates: Start 2022-04-29 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the Validity of Remote Diagnosis for Autism Spectrum Disorder in Children Aged 24 to 60 Months with Neurodevelopmental Disorders. First Test (Remote): Visit 1 - Autism Diagnostic Interview-Revised (ADI-R) | Visit 1
  The ADI-R is a structured interview conducted with parents or caregivers to assess children suspected of having Autism Spectrum Disorder (ASD). It focuses on three key areas: language/communication, social interaction, and repetitive/restrictive behaviors. The ADI-R provides a comprehensive evaluation of both current and past behaviors, and is commonly used in both clinical and research settings for diagnosis.
  Scoring:
  The ADI-R includes scores in three domains: Communication, Social Interaction, and Restricted/Repetitive Behaviors.
  Each item is scored on a scale from 0 to 3 or 0 to 9, where higher scores indicate more severe impairment.
Evaluation of the Validity of Remote Diagnosis for Autism Spectrum Disorder in Children Aged 24 to 60 Months with Neurodevelopmental Disorders. Second Test (Remote): Visit 2 - Brief Observation of Symptoms of Autism (BOSA) | Visit 2
  The BOSA is a observational tool designed to evaluate behaviors related to Autism Spectrum Disorder (ASD) in children:
  The BOSA includes scores across multiple domains: Social Affect and Restricted/Repetitive Behaviors.
  Items are typically scored on a scale from 0 to 3, where higher scores indicate more significant impairment in the observed behavior.
Standard diagnostic pathway (as usual), with the first visit conducted in person: First Test (in person): Visit 0 - Autism Diagnostic Interview-Revised (ADI-)R | Visit 0
  The ADI-R is a structured interview conducted with parents or caregivers to assess children suspected of having Autism Spectrum Disorder (ASD). It focuses on three key areas: language/communication, social interaction, and repetitive/restrictive behaviors. The ADI-R provides a comprehensive evaluation of both current and past behaviors, and is commonly used in both clinical and research settings for diagnosis.
  Scoring:
  The ADI-R includes scores in three domains: Communication, Social Interaction, and Restricted/Repetitive Behaviors.
  Each item is scored on a scale from 0 to 3 or 0 to 9, where higher scores indicate more severe impairment.
Standard diagnostic pathway (as usual), with the second visit conducted in person: Second Test (in person): Visit 3 - Autism Diagnostic Observation Schedule, Second Edition (ADOS-2): | Visit 3
  The ADOS-2 assesses two main domains: Social Affect (SA) and Restricted/Repetitive Behaviors (RRB), scored based on behavior frequency and intensity.
  The study uses three ADOS-2 modules tailored to different developmental and language levels:
  Module Toddler: For children (12-30 months) with little or no spoken language. Focuses on early social communication.
  Scores: 0 to 24. Module 1: For children over 31 months with little or no spoken language. Assesses non-verbal communication, play, and social interaction.
  Scores: 0 to 24. Module 2: For individuals using simple phrases. Focuses on verbal communication, socialization, and repetitive behaviors.
  Scores: 0 to 24 for SA, 0 to 10 for RRB. The total score combines both domains, with higher scores indicating greater impairment.
The primary objective of the study will be to assess the concordance between the gold standard in-person diagnosis and the remote diagnosis, to determine whether remote evaluations provide reliable diagnostic outcomes. | End of study (22 weeks after inclusion for all participants).
  The evaluation criteria will focus on the level of concordance between the in-person (gold standard) and remote diagnoses, using Cohen's kappa coefficient to measure agreement between the two methods.

SECONDARY OUTCOMES:
Sensitivity and Specificity of the Remote Autism Diagnostic Interview-Revised (ADI-R) in Diagnosing Autism Spectrum Disorder (ASD) | End of study (22 weeks after inclusion for all participants).
  Outcome Measure: Number of participants correctly identified with ASD (sensitivity) and number of participants correctly identified without ASD (specificity) using the remote administration of the ADI-R in comparison to the in-person diagnostic standard.
Concordance Between In-Person and Remote Autism Diagnostic Interview-Revised (ADI-R) Results" | End of study (22 weeks after inclusion for all participants).
  Outcome Measure: Agreement between in-person and remote Autism Diagnostic Interview-Revised (ADI-R) scores across all four diagnostic domains, measured using Cohen's kappa coefficient.
Concordance Between Remote Brief Observation of Symptoms of Autism (BOSA) and In-Person Autism Diagnostic Observation Schedule, Second Edition (ADOS-2) Diagnoses" | End of study (22 weeks after inclusion for all participants).
  Outcome Measure: Agreement between remote Brief Observation of Symptoms of Autism (BOSA) and in-person Autism Diagnostic Observation Schedule, Second Edition (ADOS-2) diagnoses, measured using Cohen's kappa coefficient.
Sensitivity and Specificity of the Brief Observation of Symptoms of Autism (BOSA) Compared to the Gold Standard Autism Diagnostic Observation Schedule, Second Edition (ADOS-2)" | End of study (22 weeks after inclusion for all participants).
  Outcome Measure: Sensitivity (number of participants correctly identified with Autism Spectrum Disorder) and specificity (number of participants correctly identified without Autism Spectrum Disorder) of the Brief Observation of Symptoms of Autism (BOSA) compared to the gold standard Autism Diagnostic Observation Schedule, Second Edition (ADOS-2).

CONTACTS AND LOCATIONS:
Locations (1):
- GHU Paris Psychiatrie et Neurosciences, Paris, France

IPD SHARING:
Plan to Share IPD: No